CLINICAL TRIAL: NCT04760678
Title: Clinical Aspects, Severity, Management and Outcome of Febrile Illnesses in the Democratic Republic Congo (DRC).
Brief Title: Febrile Illness in Kinshasa and Kimpese
Acronym: FIKI²
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other)
Responsible Party: Sponsor
Other Study IDs: FIKI²
Record Dates: First submitted 2021-02-12; First posted 2021-02-18 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Febrile Illness
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — No intervention (observational study in human participants)

SUMMARY:
This is a bi-centric prospective observational cohort study of adults and children presenting to the emergency room or outpatient department with community febrile illness (with or without signs of focalization) in 2 clinical sites (hospitals) in the DRC. The study will describe the epidemiology, clinical aspects, severity, management and outcome of febrile illnesses using data collected during routine diagnostic and therapeutic procedures.

Each patient will be followed for 21 days. The follow-up will include

* Daily visits for hospitalized patients,
* Telephone calls (or study center visit or home visit) on days 7, 14 and 21 for outpatients and discharged patients.

The study has been amended (EC UZA approval in June 2021) to perform a set of laboratory analyses in the partners institutions and at the ITM. We aim as a new primary objective at describing the profile of different biomarkers (C-reactive protein and white blood cell count with differentiation) in participants enrolled with febrile illness, and as secondary objectives to correlate them with outcome (assessed at day 21) and with several etiological diagnoses, especially malaria (as assessed by rapid diagnostic test and blood smear). The purpose is to investigate the potential diagnostic and prognostic value of these biomarkers which are increasingly available at the point-of-care.

ELIGIBILITY:
Inclusion Criteria:

1. Ongoing and objectified fever at presentation, or documented at home or other health center within 24 hours prior to presentation, defined by:

   * Axillary or tympanic temperature > 37.5°C OR
   * Oral or rectal temperature > 38°C
2. Possibility of contact between the patient (or designated relative) and the study team on days 7, 14 and 21
3. Informed consent signed by the patient (adults) or a legally acceptable representative (children or patients whose condition does not allow them to sign informed consent), with the consent of children as young as 12 years of age, whenever possible.

Exclusion Criteria:

1. Children less than two months old
2. Hospitalization > 48 h in the last 14 days (to exclude nosocomial fevers)

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children presenting to emergency or outpatient departments with community febrile illness (with or without signs of focus) in 2 clinical sites (hospitals) in the DRC.
Sampling Method: Probability Sample
Enrollment: 1046 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bottieau, MD, Principal Investigator — Institute of Tropical Medicine
Locations (2):
- Democratic Republic of the Congo (2):
  - IME Kimpese, Kimpese, Bas-Congo Province
  - Hôpital General de Kinshasa, Kinshasa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hauner A, Lusala SM, Roge S, Van Reet N, Cnops L, Da Luz RI, Van Esbroeck M, Kapandji M, Kuamfumu MM, Kiabanzawoko O, Phanzu DM, Verle P, Ahuka-Mundeke S, Arien KK. Development and validation of a sample-to-result real time multiplex RT-PCR test for human African trypanosomiasis and arboviral febrile illnesses in the Democratic Republic of the Congo. BMC Infect Dis. 2026 Feb 5. doi: 10.1186/s12879-026-12550-0. Online ahead of print. PMID 41645098

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: all adults and children presenting to emergency departments or outpatient clinic with community-acquired febrile illness (HGKinshasa children, HGRKimpese adults, HGR Kimpese children)
Period: Overall Study
Arm/Group | All Participants
Started | 1046
Completed | 984
Not Completed | 62
Not completed — Death | 13
Not completed — Lost to Follow-up | 48
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 997
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 5 [2 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 467
  Male | 530
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 997
Education [Count of Participants; unit: Participants]
  None | 2
  Child going to school | 468
  Missing | 413
  primary | 1
  secondary | 58
  superior | 50
  unknown | 5
Temperature [Mean (Inter-Quartile Range); unit: degrees celcius] | 37.8 [36.7 to 38.6]
Height [Mean (Inter-Quartile Range); unit: cm] | 118 [92 to 152]
Weight [Mean (Inter-Quartile Range); unit: kg] | 19 [12.5 to 35]
Brachial Perimeter [Mean (Inter-Quartile Range); unit: cm] | 15 [14 to 16]
Diastolic blood pressure [Mean (Inter-Quartile Range); unit: mm Hg] | 70 [60 to 80]
Syst. Blood pressure [Mean (Inter-Quartile Range); unit: mm Hg] | 108 [100 to 120]
Heart rate [Mean (Inter-Quartile Range); unit: BPM] | 108 [95 to 122]
Breathing rate [Mean (Inter-Quartile Range); unit: breaths per minute] | 28 [22 to 32]
SpO2 [Mean (Inter-Quartile Range); unit: %] | 98 [97 to 99]
Previous consultation [Count of Participants; unit: Participants]
  both | 7
  formal system | 72
  informal system | 11
  neither | 907
Previous treatment [Count of Participants; unit: Participants]
  yes | 875
  no | 113
  unknown | 9
Antimalarial [Count of Participants; unit: Participants]
  no | 843
  yes | 154
Antibiotic [Count of Participants; unit: Participants]
  no | 873
  yes | 124
Fever duration [Mean (Inter-Quartile Range); unit: days] | 3 [2 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Survival With Symptom Resolution
Description: Proportion of survival with symptom resolution assessed at day 21, of febrile illnesses
Time Frame: Day 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 977
percentage of participants | 96.9 [95.6 to 97.8]

2. Primary Outcome: CRP Values
Description: CRP values at day 0 (inclusion)
Time Frame: Day 0
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | All Participants
Number analyzed (Participants) | 997
mg/L | 20 [6 to 77.25]

3. Primary Outcome: White Blood Cell Count
Description: white blood cell count with differentiation at day 0 (inclusion)
Time Frame: day 0
Measure: Median (Inter-Quartile Range); unit: 10^9 cells/L
Arm/Group | All Participants
Number analyzed (Participants) | 997
10^9 cells/L | 7 [5.1 to 9.7]

4. Secondary Outcome: Proportion of Survival With Symptom Resolution
Description: Proportion of survival with symptom resolution assessed at day 7, of febrile illnesses
Time Frame: Day 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 970
percentage of participants | 93.9 [92.2 to 95.3]

5. Secondary Outcome: Proportion of Survival Without Symptom Resolution
Description: Proportion of survival without symptom resolution assessed at day 7, of febrile illnesses
Time Frame: Day 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 970
percentage of participants | 5.2 [3.9 to 6.7]

6. Secondary Outcome: Proportion of Death
Description: Proportion of death assessed at day 7, of febrile illnesses
Time Frame: Day 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 970
percentage of participants | 0.9 [0.5 to 1.8]

7. Secondary Outcome: Proportion of Survival With Symptom Resolution
Description: Proportion of survival with symptom resolution assessed at day 14, in febrile illnesses
Time Frame: Day 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 977
percentage of participants | 95.7 [94.2 to 96.8]

8. Secondary Outcome: Proportion of Survival Without Symptom Resolution
Description: Proportion of survival without symptom resolution assessed at day 14, in febrile illnesses
Time Frame: Day 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 977
percentage of participants | 3.2 [2.2 to 4.5]

9. Secondary Outcome: Proportion of Death
Description: Proportion of death assessed at day 14, in febrile ilnesses
Time Frame: Day 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 977
percentage of participants | 1.1 [0.6 to 2]

10. Secondary Outcome: Proportion of Survival Without Symptom Resolution
Description: Proportion of survival without symptom resolution assessed at day 21, in febrile illnesses
Time Frame: Day 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 997
percentage of participants | 1.8 [1.1 to 2.8]

11. Secondary Outcome: Proportion of Death
Description: Proportion of death assessed at day 21, in febrile illnesses
Time Frame: Day 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 997
percentage of participants | 1.3 [0.8 to 2.2]

12. Secondary Outcome: Proportion of Participants With Initial Hospitalization
Description: Proportion of participants with initial hospitalization (assessed at Day 21)
Time Frame: Day 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 997
percentage of participants | 13.3 [11.4 to 15.6]

13. Secondary Outcome: Proportion of Participants With Secondary Hospitalization
Description: Proportion of participants with secondary hospitalization assessed at day 21
Time Frame: Day 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 997
percentage of participants | 1.1 [0.6 to 2]

14. Secondary Outcome: Length of Hospital Stay (Initial and/or Secondary Hospitalization)
Description: Length of hospital stay (initial and/or secondary hospitalization) assessed at day 21
Time Frame: Day 21
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 997
days | 5 [3 to 8]

15. Secondary Outcome: Number of Secondary Visits
Description: Number of secondary visits (assessed at Day 21).
Time Frame: Day 21
Measure: Median (Inter-Quartile Range); unit: visits
Arm/Group | All Participants
Number analyzed (Participants) | 997
visits | 4 [4 to 4]

16. Secondary Outcome: Patient Outcomes
Description: Association of CRP values and white blood cell counts with patient outcomes
Time Frame: Day 21
Population: overal number of pts analyzed = number resolved + number non resolved
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | All Participants
Number analyzed (Participants) | 984
mg/L
  CRP clinical outcome Resolution: number analyzed (Participants) | 966
  CRP clinical outcome Resolution | 19 [6 to 72]
  CRP clinical outcome Non-resolution: number analyzed (Participants) | 18
  CRP clinical outcome Non-resolution | 71 [13 to 87.5]
Statistical Analysis 1: Comparison: All Participants; Test type: Other — Fisher's exact test; p = 0.107, Fisher Exact

17. Secondary Outcome: Severity of Illness
Description: Severity of illness on day 0 as assessed by the ASAPS/IGSA (Simplified ambulatory severity index) score in adult febrile illnesses.
  IGSA is a clinical severity score designed to estimate the prognosis of patients in emergency settings. It is based on six clinical parameters: age, heart rate (pulse), systolic blood pressure, respiratory rate, body temperature, and Glasgow Coma Scale score. Each parameter is assigned a score from 0 to 4 based on the severity of the observed abnormality. The total score is the sum of the individual scores for each parameter, with a theoretical maximum of 24 points.
  The ASAPS/IGSA score can be calculated with a calculator via the website of société Française de Médecine d'urgence.
  A value between 0 and 24 is expected, it's life-threatening if ≥ 8. The lower the total score, the more favorable the prognosis.
Time Frame: Day 0
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Adults: all adults presenting to emergency departments or outpatient clinic with community-acquired febrile illness (HGRKimpese adults)
Arm/Group | Adults
Number analyzed (Participants) | 121
score on a scale | 2 [1 to 4]

18. Secondary Outcome: Severity of Illness
Description: Severity of illness on day 0 as assessed by the qSOFA (Quick Sepsis Related Organ Failure Assessment) score in adult febrile illnesses.
  qSOFA is a clinical tool to identify patients with suspected infection who are at greater risk for poor outcomes, such as in-hospital mortality or prolonged intensive care unit (ICU) stays. It is particularly useful in non-ICU settings like emergency departments.
  The qSOFA score evaluates 3 clinical criteria, assigning 1 point for each (it's the sum of 3 criteria):
  * Respiratory Rate: ≥22 breaths per minute.
  * Systolic Blood Pressure: ≤100 mmHg.
  * Altered Mental Status: Glasgow Coma Scale (GCS) score <15. Each criterion is scored as follows: 1 point for meeting the threshold of each criterion.
  The total qSOFA score ranges from 0-3 points.
  Interpretation of Scores:
  0 point: Low risk for poor outcomes
  1. point: Moderate risk; consider monitoring and reassessment
  2. or 3 points: High risk; prompt evaluation and intervention recommended
Time Frame: Day 0
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Adults
Number analyzed (Participants) | 121
score on a scale | 1 [0 to 2]

19. Secondary Outcome: Severity of Illness
Description: Severity of illness on day 7 as assessed by the ASAPS/IGSA score (Simplified ambulatory severity index score) in adult febrile illnesses.
  IGSA is a clinical severity score designed to estimate the prognosis of patients in emergency settings. It is based on six clinical parameters: age, heart rate (pulse), systolic blood pressure, respiratory rate, body temperature, and Glasgow Coma Scale score. Each parameter is assigned a score from 0 to 4 based on the severity of the observed abnormality. The total score is the sum of the individual scores for each parameter, with a theoretical maximum of 24 points.
  The ASAPS/IGSA score can be calculated with a calculator via the website of société Française de Médecine d'urgence.
  A value between 0 and 24 is expected, it's life-threatening if ≥ 8. The lower the total score, the more favorable the prognosis.
Time Frame: day 7
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Adults
Number analyzed (Participants) | 23
score on a scale | 0 [0 to 1.5]

20. Secondary Outcome: Severity of Illness
Description: Severity of illness on day 7 as assessed by the qSOFA (Quick Sepsis Related Organ Failure Assessment) score in adult febrile illnesses.
  qSOFA is a clinical tool to identify patients with suspected infection who are at greater risk for poor outcomes, such as in-hospital mortality or prolonged intensive care unit (ICU) stays. It is particularly useful in non-ICU settings like emergency departments.
  The qSOFA score evaluates 3 clinical criteria, assigning 1 point for each (it's the sum of 3 criteria):
  * Respiratory Rate: ≥22 breaths per minute.
  * Systolic Blood Pressure: ≤100 mmHg.
  * Altered Mental Status: Glasgow Coma Scale (GCS) score <15. Each criterion is scored as follows: 1 point for meeting the threshold of each criterion.
  The total qSOFA score ranges from 0-3 points.
  Interpretation of Scores:
  0 point: Low risk for poor outcomes
  1. point: Moderate risk; consider monitoring and reassessment
  2. or 3 points: High risk; prompt evaluation and intervention recommended
Time Frame: Day 7
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Adults
Number analyzed (Participants) | 23
score on a scale | 1 [0 to 1]

21. Secondary Outcome: Severity of Illness
Description: Severity of illness on day 14 as assessed by the ASAPS/IGSA (Simplified ambulatory severity index) score in adult febrile illnesses.
  IGSA is a clinical severity score designed to estimate the prognosis of patients in emergency settings. It is based on six clinical parameters: age, heart rate (pulse), systolic blood pressure, respiratory rate, body temperature, and Glasgow Coma Scale score. Each parameter is assigned a score from 0 to 4 based on the severity of the observed abnormality. The total score is the sum of the individual scores for each parameter, with a theoretical maximum of 24 points.
  The ASAPS/IGSA score can be calculated with a calculator via the website of société Française de Médecine d'urgence.
  A value between 0 and 24 is expected, it's life-threatening if ≥ 8. The lower the total score, the more favorable the prognosis.
Time Frame: Day 14
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Adults
Number analyzed (Participants) | 12
score on a scale | 1.5 [0 to 2.25]

22. Secondary Outcome: Severity of Illness
Description: Severity of illness on day 14 as assessed by the qSOFA (Quick Sepsis Related Organ Failure Assessment) score in adult febrile illnesses.
  qSOFA is a clinical tool to identify patients with suspected infection who are at greater risk for poor outcomes, such as in-hospital mortality or prolonged intensive care unit (ICU) stays. It is particularly useful in non-ICU settings like emergency departments.
  The qSOFA score evaluates 3 clinical criteria, assigning 1 point for each (it's the sum of 3 criteria):
  * Respiratory Rate: ≥22 breaths per minute.
  * Systolic Blood Pressure: ≤100 mmHg.
  * Altered Mental Status: Glasgow Coma Scale (GCS) score <15. Each criterion is scored as follows: 1 point for meeting the threshold of each criterion.
  The total qSOFA score ranges from 0-3 points.
  Interpretation of Scores:
  0 point: Low risk for poor outcomes
  1. point: Moderate risk; consider monitoring and reassessment
  2. or 3 points: High risk; prompt evaluation and intervention recommended
Time Frame: Day 14
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Adults
Number analyzed (Participants) | 12
score on a scale | 1 [0 to 1]

23. Secondary Outcome: Severity of Illness
Description: Severity of illness on day 21 as assessed by the ASAPS/IGSA (Simplified ambulatory severity index) score in adult febrile illnesses.
  IGSA is a clinical severity score designed to estimate the prognosis of patients in emergency settings. It is based on six clinical parameters: age, heart rate (pulse), systolic blood pressure, respiratory rate, body temperature, and Glasgow Coma Scale score. Each parameter is assigned a score from 0 to 4 based on the severity of the observed abnormality. The total score is the sum of the individual scores for each parameter, with a theoretical maximum of 24 points.
  The ASAPS/IGSA score can be calculated with a calculator via the website of société Française de Médecine d'urgence.
  A value between 0 and 24 is expected, it's life-threatening if ≥ 8. The lower the total score, the more favorable the prognosis.
Time Frame: Day 21
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Adults
Number analyzed (Participants) | 17
score on a scale | 1 [0 to 2]

24. Secondary Outcome: Severity of Illness
Description: Severity of illness on day 21 as assessed by the qSOFA (Quick Sepsis Related Organ Failure Assessment)score in adult febrile illnesses.
  qSOFA is a clinical tool to identify patients with suspected infection who are at greater risk for poor outcomes, such as in-hospital mortality or prolonged intensive care unit (ICU) stays. It is particularly useful in non-ICU settings like emergency departments.
  The qSOFA score evaluates 3 clinical criteria, assigning 1 point for each (it's the sum of 3 criteria):
  * Respiratory Rate: ≥22 breaths per minute.
  * Systolic Blood Pressure: ≤100 mmHg.
  * Altered Mental Status: Glasgow Coma Scale (GCS) score <15. Each criterion is scored as follows: 1 point for meeting the threshold of each criterion.
  The total qSOFA score ranges from 0-3 points.
  Interpretation of Scores:
  0 point: Low risk for poor outcomes
  1. point: Moderate risk; consider monitoring and reassessment
  2. or 3 points: High risk; prompt evaluation and intervention recommended
Time Frame: Day 21
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Adults
Number analyzed (Participants) | 17
score on a scale | 1 [0 to 1]

25. Secondary Outcome: Frequency of Malaria
Description: Frequency of malaria as detected by rapid test (HRP II antigen) at day 21 in febrile illnesses
Time Frame: Day 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 774
percentage of participants | 31.6 [28.3 to 35]

26. Secondary Outcome: Frequency of Malaria
Description: Frequency of malaria as detected by rapid test (pLDH antigen) at day 21 in febrile illnesses
Time Frame: Day 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 774
percentage of participants | 22.3 [19.5 to 25.4]

27. Secondary Outcome: Frequency of Malaria
Description: Frequency of malaria as detected by thick smear positivity at day 21 in febrile illnesses
Time Frame: Day 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 790
percentage of participants | 25.3 [22.3 to 28.6]

28. Secondary Outcome: Frequency of Malaria
Description: Frequency of malaria type Plasmodium falciparum as detected by thick smear at day 21
Time Frame: Day 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 790
percentage of participants | 24.3 [21.4 to 27.5]

29. Secondary Outcome: Parasitemia of Malaria
Description: Parasitemia as detected by thick smear at day 21 in febrile illnesses
Time Frame: Day 21
Measure: Median (Inter-Quartile Range); unit: trophozoïtes/microliter
Arm/Group | All Participants
Number analyzed (Participants) | 790
trophozoïtes/microliter | 8350 [1924 to 41892]

30. Secondary Outcome: Frequency of Malaria
Description: Frequency of malaria type Plasmodium malariae as detected by thick smear at day 21
Time Frame: Day 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 790
percentage of participants | 1.1 [0.5 to 2.1]

ADVERSE EVENTS:
Time Frame: All cause mortality was collected over 21 days. No adverse event data collected as no study medication administered.
Description: No medication administered in the study so no adverse event data collection
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 13/997
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT04760678/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT04760678/SAP_001.pdf